CLINICAL TRIAL: NCT03965533
Title: A Randomised, Double-blind, Placebo-controlled Phase I Study of the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Intravenous Dose of GSK2831781 in Healthy Japanese and Caucasian Participants, and a Single Subcutaneous Dose of GSK2831781 in Healthy Caucasian Participants
Brief Title: Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of GSK2831781 After an Intravenous (IV) Dose in Healthy Japanese and Caucasian Subjects, and a Subcutaneous (SC) Dose in Healthy Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207823
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
Keywords: Japanese, Caucasian, pharmacokinetics, pharmacodynamics, GSK2831781, lymphocyte activation gene-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Placebo IV- Caucasian Participants (Placebo Comparator): Caucasian male participants were administered a single IV infusion of 0.9% weight by volume (w/v) saline placebo.
  Interventions: Drug: Placebo
- Part A: GSK2831781 450 mg IV- Caucasian Participants (Experimental): Caucasian male participants were administered a single IV infusion of GSK2831781 at a dose of 450 milligram (mg), diluted in 0.9% w/v saline.
  Interventions: Drug: GSK2831781
- Part A: Placebo IV- Japanese Participants (Placebo Comparator): Japanese male participants were administered a single IV infusion of 0.9% w/v saline placebo.
  Interventions: Drug: Placebo
- Part A: GSK2831781 450 mg IV- Japanese Participants (Experimental): Japanese male participants were administered a single IV infusion of GSK2831781 at a dose of 450 mg, diluted in 0.9% w/v saline.
  Interventions: Drug: GSK2831781
- Part B: Placebo SC (Placebo Comparator): Caucasian male participants were administered three SC injections of 0.9% w/v saline placebo.
  Interventions: Drug: Placebo
- Part B: GSK2831781 150 mg SC (Experimental): Caucasian male participants were administered a single SC injection of a unit dose strength of 150 mg per milliliter (mL) of GSK2831781, diluted in 0.9% w/v saline. Participants also received 2 dummy injections of 0.9% w/v saline placebo SC to maintain the blinding.
  Interventions: Drug: GSK2831781
- Part B: GSK2831781 450 mg SC (Experimental): Caucasian male participants were administered three SC injections of a unit dose strength of 150 mg per mL of GSK2831781 to achieve a dose of 450 mg.
  Interventions: Drug: GSK2831781

INTERVENTIONS:
Drug: GSK2831781 — GSK2831781 will be available as Dose-1 and Dose-2 as IV infusion or SC injection. Subjects will receive GSK2831781 Dose-1 IV diluted in 0.9% saline or GSK2831781 SC as multiples of Dose-2 SC.
  Arms: Part A: GSK2831781 450 mg IV- Caucasian Participants; Part A: GSK2831781 450 mg IV- Japanese Participants; Part B: GSK2831781 150 mg SC; Part B: GSK2831781 450 mg SC
Drug: Placebo — Placebo will be 0.9% saline solution which will be administered in subjects as IV infusion or SC injection.
  Arms: Part A: Placebo IV- Caucasian Participants; Part A: Placebo IV- Japanese Participants; Part B: Placebo SC

SUMMARY:
This is a double-blind, placebo-controlled, randomized, parallel group, two-part study where single IV doses of GSK2831781 will be administered to healthy Japanese and Caucasian subjects in part A and SC doses will be administered to healthy Caucasian subjects in part B. GSK2831781 is a humanized, antibody-dependent cell cytotoxicity (ADCC) enhanced depleting monoclonal antibody that is specific to the lymphocyte activation gene-3 (LAG3) protein. LAG3 is a transmembrane receptor, which is upregulated on T cells following activation. The objective of the study is to assess the safety, tolerability, PK, PD and immunogenicity post administration of GSK2831781 in healthy subjects. The duration of the study is approximately 147 days for each subject enrolled. Approximately 36 subjects will be enrolled in the study, 16 subjects in Part A and 20 subjects in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12-lead ECGs. A subject with a clinical abnormality or laboratory parameter(s) outside the reference range for the population being studied that is not specifically listed in the inclusion or exclusion criteria may be included if the Investigator (in consultation with the Medical Monitor if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or interpretation.
* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight >=40 kilogram (kg) and body mass index (BMI) <=30 kilogram per meter square (kg/m^2).
* Male.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Japanese ancestry, defined as having been born in Japan, being descendants of four ethnic Japanese grandparents and two ethnic Japanese parents, holding a Japanese passport or identity papers, and being able to speak Japanese. Subjects should have lived outside Japan for less than 10 years at the time of screening.
* Caucasian ancestry, defined as Caucasian descent as evidenced by appearance and verbal confirmation of familial heritage (a subject has 2 Caucasian parents and 4 Caucasian grandparents).

Exclusion Criteria:

* History or presence of a disease that in the opinion of the investigator constitutes a risk when taking the study intervention or interfering with study assessment or interpretation of the data.
* A medical history of severe allergic reaction, angioedema, anaphylaxis, clinically significant drug hypersensitivity reaction, or autoimmune or immunodeficiency disorder.
* An active infection or a history of serious infections as follows:

  1. Use of antimicrobials (antibacterials, antivirals, antifungals or antiparasitic agents) for an infection within 30 days before first dose. Topical treatments may be allowed at the Medical Monitor's discretion.
  2. A history of opportunistic infections.
  3. Recurrent or chronic infection, or other active infection, that in the opinion of the Investigator might cause this study to be detrimental to the subject.
  4. Symptomatic herpes zoster within 3 months prior to screening.
  5. History of tuberculosis (TB) (active or latent) irrespective of treatment status.
  6. A positive diagnostic TB test at screening (defined as a positive QuantiFERON test). In cases where the QuantiFERON test is indeterminate, the subject may have the test repeated once and if their second test is negative they will be eligible. In the event a second test is also indeterminate, the investigator has the option to undertake purified protein derivative (PPD) testing. If the PPD reaction is <5 millimeter (mm) at 48 to 72 hours, then the subject is eligible. If the reaction is >=5 mm, or PPD testing is not undertaken, the subject is not eligible.
* Any planned major surgical procedure during the study.
* A history of malignant neoplasm within the last 10 years, except for fully treated nonmetastatic basal or squamous cell cancers of the skin (within 3 years) that shows no evidence of recurrence.
* Use of prescription or non-prescription drugs (including recreational drugs and herbal medications) within 7 days or 5 half-lives (whichever is longer) prior to dosing, unless in the opinion of the investigator, the medication will not interfere with the study or compromise subject safety. Paracetamol (acetaminophen) at doses of <=4 grams per day, and occasional use of non-steroidal anti-inflammatory drugs (NSAIDs) at licensed doses, are permitted.
* Received live vaccination within 4 weeks of Day 1, or plan to receive a live vaccination during the study until follow-up.
* Previous exposure to GSK2831781, or hypersensitivity to any excipients in the clinical formulation of GSK2831781.
* Treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Participation in a clinical trial and has received an investigational medicinal product (IMP) within the following time period prior to screening in the current study: 3 months, 5 half-lives, or twice the duration of the biological effect of the IMP (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* Neutrophil or lymphocyte counts below the normal range.
* eGFR by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation <=90 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) at screening.
* ALT >2x upper limit of normal (ULN) and bilirubin >1.5x ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* Other clinically significant abnormalities of laboratory assessments, as judged by the Investigator and/or GSK Medical Monitor, that could affect the safety of the subject, or the interpretation of the data from the study.
* Presence of hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb), or positive hepatitis C antibody result at screening (Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled only if a confirmatory negative Hepatitis C ribonucleic acid [RNA] test is obtained).
* Positive serology for human immunodeficiency virus (HIV) at screening.
* Positive pre-study drug/alcohol screen.
* QTc >450 millisecond (msec), based on the mean of triplicate ECGs. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF; preferred method), or another method, machine or overread.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 grams (g) of alcohol: a halfpint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Unstable lifestyle factors, to the extent that in the opinion of the investigator they would interfere with the ability of a subject to complete the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subjects will be included in the study
Enrollment: 36 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, placebo-controlled, randomized, parallel group, two-part study to evaluate safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of intravenous (IV) dose of GSK2831781 in healthy Japanese and Caucasian participants (Part A) and subcutaneous (SC) dose of GSK2831781 in healthy Caucasian participants (Part B).
Pre-assignment Details: A total of 30 participants were screened and 16 participants were enrolled in Part A (14 were screen failures). A total of 41 participants were screened and 20 participants were enrolled in Part B (21 were screen failures). Placebo arms across similar dosing strategies were combined in Part B.
Groups:
- Part B: GSK2831781 150 mg SC: Arm Description: Caucasian male participants were administered a single SC injection of a unit dose strength of 150 mg per milliliter (mL) of GSK2831781, diluted in 0.9% w/v saline. Participants also received 2 dummy injections of 0.9% w/v saline placebo SC to maintain the blinding.
Period: Part A (112 Days)
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Started | 2 | 6 | 2 | 6 | 0 | 0 | 0
Completed | 2 | 6 | 2 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (112 Days)
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Started | 0 | 0 | 0 | 0 | 4 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 4 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC | Total
Number analyzed (Participants) | 2 | 6 | 2 | 6 | 4 | 8 | 8 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 2 | 6 | 4 | 8 | 8 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 6 | 2 | 6 | 4 | 8 | 8 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-White/Caucasian/European Heritage (H) | 2 | 6 | 0 | 0 | 4 | 8 | 8 | 28
  Asian-Japanese H/East Asian H/South East Asian H | 0 | 0 | 2 | 6 | 0 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician. Number of participants who had SAEs and non-SAEs are presented.
Time Frame: Up to Day 112
Population: Safety Population comprised of all randomized (all participants who were randomized into the study and received a randomization number) participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants
  Non-SAEs | 2 | 5 | 0 | 4
  SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician. Number of participants who had SAEs and non-SAEs are presented.
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants
  Non-SAEs | 4 | 6 | 4
  SAEs | 0 | 1 | 0

3. Primary Outcome: Part A: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital signs were measured in a semi-supine position after five minutes of rest and included temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate. The clinical concern range for the parameters were: SBP (low: <85 millimeters of mercury [mmHg] and high: >160 mmHg), DBP (low: <45 mmHg and high: >100 mmHg), heart rate (low: <40 beats per minute [bpm] and high: >110 bpm) and temperature (low: <35 degrees celsius [°C] and high: >=37.5 °C). Number of participants with any vital sign value of potential clinical importance is reported.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants | 0 | 1 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital signs were measured in a semi-supine position after five minutes of rest and included temperature, SBP, DBP and heart rate. The clinical concern range for the parameters were: SBP (low: <85 mmHg and high: >160 mmHg), DBP (low: <45 mmHg and high: >100 mmHg), heart rate (low: <40 bpm and high: >110 bpm) and temperature (low: <35 °C and high: >=37.5 °C). Number of participants with any vital sign value of potential clinical importance is reported.
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants | 1 | 0 | 1

5. Primary Outcome: Part A: Number of Participants With Any Hematology Parameter of Potential Clinical Importance
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (high: >0.54 proportion of red blood cells in blood and low: change from Baseline <0.075 proportion of red cells in blood); hemoglobin (high: >180 grams per liter [g/L] and low: change from Baseline <25 g/L), lymphocytes (low: <0.8 Giga cells per liter [Giga cells/L]); neutrophil count (low: <1.5 Giga cells/L); eosinophil count (high: >1 Giga cells/L); platelet count (low: <100 Giga cells/L and high: >550 Giga cells/L) and white blood cells count (low: <3 Giga cells/L and high: >20 Giga cells/L). Number of participants with any hematology parameter value of potential clinical importance is reported.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants | 0 | 1 | 0 | 2

6. Primary Outcome: Part B: Number of Participants With Any Hematology Parameter of Potential Clinical Importance
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (high: >0.54 proportion of red blood cells in blood and low: change from Baseline <0.075 proportion of red cells in blood); hemoglobin (high: >180 g/L and low: change from Baseline <25 g/L), lymphocytes (low: <0.8 Giga cells/L); neutrophil count (low: <1.5 Giga cells/L); eosinophil count (high: >1 Giga cells/L); platelet count (low: <100 Giga cells/L and high: >550 Giga cells/L) and white blood cells count (low: <3 Giga cells/L and high: >20 Giga cells/L). Number of participants with any hematology parameter value of potential clinical importance is reported.
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants | 0 | 0 | 1

7. Primary Outcome: Part A: Number of Participants With Any Clinical Chemistry Parameter of Potential Clinical Importance
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: alanine aminotransferase (high: >=2 times upper limit of normal [ULN]); aspartate aminotransferase (high: >=2 times ULN); alkaline phosphatase (high: >=2 times ULN); total bilirubin (high: >=1.5 times ULN); blood urea nitrogen (high: >10.5 millimoles per liter [mmol/L]); calcium (low: <2 mmol/L and high: >2.75 mmol/L); creatinine (high: change from Baseline >26 micromoles per liter); estimated glomerular filtration rate (low: <60 milliliter per minute per 1.73 squared meter); glucose (low: <3 mmol/L and high: >9 mmol/L); potassium (low: <3 mmol/L and high: >5.5 mmol/L); sodium (low: <130 mmol/L and high: >150 mmol/L) and total protein (low: <50 g/L and high: >85 g/L). Number of participants with any clinical chemistry parameter value of potential clinical importance is reported.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 1

8. Primary Outcome: Part B: Number of Participants With Any Clinical Chemistry Parameter of Potential Clinical Importance
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: alanine aminotransferase (high: >=2 times ULN); aspartate aminotransferase (high: >=2 times ULN); alkaline phosphatase (high: >=2 times ULN); total bilirubin (high: >=1.5 times ULN); blood urea nitrogen (high: >10.5 mmol/L]); calcium (low: <2 mmol/L and high: >2.75 mmol/L); creatinine (high: change from Baseline >26 micromoles per liter); estimated glomerular filtration rate (low: <60 milliliter per minute per 1.73 squared meter); glucose (low: <3 mmol/L and high: >9 mmol/L); potassium (low: <3 mmol/L and high: >5.5 mmol/L); sodium (low: <130 mmol/L and high: >150 mmol/L) and total protein (low: <50 g/L and high: >85 g/L). Number of participants with any clinical chemistry parameter value of potential clinical importance is reported.
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants | 0 | 0 | 1

9. Primary Outcome: Part A: Number of Participants With Any Urinalysis Parameter of Potential Clinical Importance (PCI)
Description: Urine samples were analyzed for bilirubin (Bil.),glucose (Gl.),ketones (Keto),leukocytes (leuko),nitrite (Nit.),occult blood (OB) and protein (Pro.) by dipstick method. Urine red blood cells (RBC) and white blood cells (WBC) were assessed by microscopy. Urine potential of hydrogen (pH) and specific gravity (Sp.Gr.) were also analyzed. The dipstick results are read as Trace,1+,2+ indicating proportional concentrations. pH is measured on a numeric scale of 0 to 14 (pH 7: neutral, pH <7: acidic and pH >7: basic). Urine Sp. Gr. is a measure of the concentration of solutes in the urine and indicated as ratio of urine density to water density. The clinical concern range for these parameters were: Bil., Gl., Leuko, OB and Pro. (high: >1+),Keto (high: >2+),Nit. (high: positive),pH (low: <4.6 and high: >8),Sp.Gr. (low: <1.001 and high: >1.035),RBC (high: >3 cells/high power field [hpf]) and WBC (high: >5 cells/hpf). Number of participants with any urinalysis parameter value of PCI is reported.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants | 2 | 0 | 0 | 1

10. Primary Outcome: Part B: Number of Participants With Any Urinalysis Parameter of Potential Clinical Importance
Description: Urine samples were analyzed for Bil., Gl., Keto, leuko, Nit., OB and Pro. by dipstick method. Urine RBC and WBC were assessed by microscopy. Urine pH and Sp.Gr. were also analyzed. The dipstick results are read as Trace, 1+, 2+ indicating proportional concentrations. pH is measured on a numeric scale of 0 to 14 (pH 7: neutral, pH <7: acidic and pH >7: basic). Urine Sp. Gr. is a measure of the concentration of solutes in the urine and indicated as ratio of urine density to water density. The clinical concern range for these parameters were: Bil., Gl., Leuko, OB and Pro. (high: >1+), Keto (high: >2+), Nit. (high: positive), pH (low: <4.6 and high: >8), Sp.Gr. (low: <1.001 and high: >1.035), RBC (high: >3 cells/hpf) and WBC (high: >5 cells/hpf). Number of participants with any urinalysis parameter value of PCI is reported.
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants | 1 | 0 | 0

11. Primary Outcome: Part A: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were recorded with the participants in a semi-supine position, after 5 minutes of rest using an ECG machine that automatically calculated heart rate and measured PR, QRS, QT and corrected QT (QTc) intervals. Number of participants with worst-case clinically significant and not clinically significant abnormal ECG findings have been presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants
  Abnormal-not Clinically significant | 1 | 0 | 0 | 0
  Abnormal-Clinically significant | 0 | 0 | 0 | 0

12. Primary Outcome: Part B: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were recorded with the participants in a semi-supine position, after 5 minutes of rest using an ECG machine that automatically calculated heart rate and measured PR, QRS, QT and QTc intervals. Number of participants with worst-case clinically significant and not clinically significant abnormal ECG findings have been presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants
  Abnormal-not Clinically significant | 0 | 1 | 0
  Abnormal-Clinically significant | 0 | 0 | 0

13. Primary Outcome: Part A: Number of Participants With Injection Site Reaction
Description: Local tolerability as measured by injection site reaction example; bruise at the site of injection and/or itching, pain, blistering or skin damage. Number of participants with any injection site reaction are presented.
Time Frame: Up to 24 hours (Day 1)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 2

14. Primary Outcome: Part B: Number of Participants With Injection Site Reaction
Description: as for outcome 13
Time Frame: Up to Day 8
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants | 0 | 0 | 0

15. Secondary Outcome: Part A: Area Under the Plasma Drug Concentration Versus Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC[0 to t]) of GSK2831781 Following IV Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1 (Pre-dose and 1, 2, 6, 12, 24 hours post-dose); Days 3, 4, 8, 15, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population comprised of all safety participants for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 6 | 6
Hours*micrograms per milliliter | 44261.755 (23.8009) | 49650.933 (19.6053)

16. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of GSK2831781 Following IV Dose
Description: as for outcome 15
Time Frame: Day 1 (Pre-dose and 1, 2, 6, 12, 24 hours post-dose); Days 3, 4, 8, 15, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 6 | 6
Micrograms per milliliter | 137.61 (22.449) | 166.20 (20.428)

17. Secondary Outcome: Part A: Time to Maximum Observed Plasma Concentration (Tmax) of GSK2831781 Following IV Dose
Description: as for outcome 15
Time Frame: Day 1 (Pre-dose and 1, 2, 6, 12, 24 hours post-dose); Days 3, 4, 8, 15, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 6 | 6
Hours | 1.980 [1.98 to 2.17] | 1.990 [1.95 to 6.02]

18. Secondary Outcome: Part B: AUC(0 to t) of GSK2831781 Following SC Dose
Description: as for outcome 15
Time Frame: Day 1 (Pre-dose); Days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 8 | 8
Hours*micrograms per milliliter | 6633.227 (26.6369) | 24269.036 (40.4247)

19. Secondary Outcome: Part B: Cmax of GSK2831781 Following SC Dose
Description: as for outcome 15
Time Frame: Day 1 (Pre-dose); Days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 8 | 8
Micrograms per milliliter | 14.61 (30.229) | 41.13 (34.252)

20. Secondary Outcome: Part B: Tmax of GSK2831781 Following SC Dose
Description: as for outcome 15
Time Frame: Day 1 (Pre-dose); Days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 8 | 8
Hours | 95.750 [46.92 to 167.75] | 120.270 [69.72 to 169.73]

21. Secondary Outcome: Part A and Part B: Bioavailability (F) of GSK2831781 Following IV Dosing at 450 mg (Caucasian and Japanese Participants) or SC Dosing at 150 mg and 450 mg (Caucasian Participants)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis in Part A (IV dose) and Part B (SC doses). Bioavailability of GSK2831781 was estimated by fitting a population pharmacokinetic model to all available data (Part A and Part B) of GSK2831781 concentrations in plasma and total soluble lymphocyte activation gene-3 (LAG3) concentrations in serum and was expressed as a percentage.
Time Frame: Part A (IV): Day 1 (Pre-dose and 1, 2, 6, 12, 24 hours post-dose); Days 3, 4, 8, 15, 22, 29, 43, 57, 71, 85 and 112; Part B (SC): Day 1 (Pre-dose); Days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 112
Population: Pharmacokinetic Population. Given the non-linearity in pharmacokinetics, a population pharmacokinetic analysis of pooled data from Part A and Part B was more appropriate. Hence, this outcome measure was estimated on pooled data from Part A and Part B.
Measure: Number (95% Confidence Interval); unit: Percentage Bioavailability
Groups:
- Part A and Part B: All Participants: In Part A, Caucasian and Japanese male participants were administered a single IV infusion of GSK2831781 at a dose of 450 mg, diluted in 0.9% w/v saline. In Part B, Caucasian male participants were administered a single SC injection of a unit dose strength of 150 mg per mL of GSK2831781, diluted in 0.9% w/v saline and also received 2 dummy injections of 0.9% w/v saline placebo SC to maintain the blinding. To achieve a dose of 450 mg, Caucasian male participants were administered three SC injections of a unit dose strength of 150 mg per mL of GSK2831781.
Arm/Group | Part A and Part B: All Participants
Number analyzed (Participants) | 28
Percentage Bioavailability | 76.5 [76.5 to 76.5]

22. Secondary Outcome: Degradation Rate of LAG3 Positive T Cells (Kout) Derived From Statistical Analysis of the Relationship Between LAG3 Positive T Cell Levels in Blood and GSK2831781 Concentrations in Plasma (Part A and Part B)
Description: Blood samples were collected to measure LAG3 positive T cell levels. Plasma samples were collected to measure concentrations of GSK2831781 in plasma. The relationship between the pharmacodynamic measure (LAG3 positive T cell levels in blood) and plasma concentrations of GSK2831781 was described by an indirect response (Emax type) pharmacokinetic/pharmacodynamic (PK/PD) model. Kout was calculated by fitting the PK/PD model to all available data (Part A and Part B) of GSK2831781 concentrations in plasma and LAG3 positive T cells in blood. The model parameter; Kout is presented.
Time Frame: Up to Day 112
Population: Pharmacokinetic Population. Given the limited dose range (150 mg-450 mg) in each part, a population PK/PD analysis of combined data from Part A and Part B was more appropriate. Hence, this outcome measure was estimated on combined data from Part A and Part B.
Measure: Mean (95% Confidence Interval); unit: Per hour
Arm/Group | Part A and Part B: All Participants
Number analyzed (Participants) | 28
Per hour | 0.0256 [0.0161 to 0.0405]

23. Secondary Outcome: Baseline of LAG3 Positive T Cell Count (CELL0) Derived From Statistical Analysis of the Relationship Between LAG3 Positive T Cell Levels in Blood and GSK2831781 Concentrations in Plasma (Part A and B)
Description: Blood samples were collected to measure LAG3 positive T cell levels. Plasma samples were collected to measure concentrations of GSK2831781 in plasma. The relationship between the pharmacodynamic measure (LAG3 positive T cell levels in blood) and plasma concentrations of GSK2831781 was described by an indirect response (Emax type) PK/PD model. CELL0 was calculated by fitting the PK/PD model to all available data (Part A and Part B) of GSK2831781 concentrations in plasma and LAG3 positive T cells in blood. The model parameter; CELL0 is presented.
Time Frame: Up to Day 112
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: Cells per microliter
Arm/Group | Part A and Part B: All Participants
Number analyzed (Participants) | 28
Cells per microliter | 1.15 [1.11 to 1.19]

24. Secondary Outcome: Concentration of Free GSK2831781 at Which Half Maximum Effect on Kout is Achieved (EC50) Derived From Statistical Analysis of the Relationship Between LAG3 Positive T Cell Levels in Blood and GSK2831781 Concentrations in Plasma (Part A and B)
Description: Blood samples were collected to measure LAG3 positive T cell levels. Plasma samples were collected to measure concentrations of GSK2831781 in plasma. The relationship between the pharmacodynamic measure (LAG3 positive T cell levels in blood) and plasma concentrations of GSK2831781 was described by an indirect response (Emax type) PK/PD model. EC50 was calculated by fitting the PK/PD model to all available data (Part A and Part B) of GSK2831781 concentrations in plasma and LAG3 positive T cells in blood. As there was a limited dose range, to allow for a successful model conversion, EC50 was fixed to the EC50 value estimated from a previous study. The model parameter; EC50 is presented.
Time Frame: Up to Day 112
Population: Pharmacokinetic Population. Given the limited dose range (150 mg-450 mg) in each part, a population PK/PD analysis of combined data from Part A and Part B was more appropriate. This outcome measure was fixed to the EC50 value estimated from a previous study.
Measure: Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | Part A and Part B: All Participants
Number analyzed (Participants) | 28
Nanograms per milliliter | 9509 [174 to 540000]

25. Secondary Outcome: Maximum Effect of Change in Kout (Emax) Derived From Statistical Analysis of the Relationship Between LAG3 Positive T Cell Levels in Blood and GSK2831781 Concentrations in Plasma (Part A and B)
Description: Blood samples were collected to measure LAG3 positive T cell levels. Plasma samples were collected to measure concentrations of GSK2831781 in plasma. The relationship between the pharmacodynamic measure (LAG3 positive T cell levels in blood) and plasma concentrations of GSK2831781 was described by an indirect response (Emax type) PK/PD model. Emax, a unitless parameter that describes the maximum change in Kout at infinite GSK2831781 concentration, was calculated by fitting the PK/PD model to all available data (Part A and Part B) of GSK2831781 concentrations in plasma and LAG3 positive T cells in blood. The model parameter; Emax is presented.
Time Frame: Up to Day 112
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Part A and Part B: All Participants
Number analyzed (Participants) | 28
Unitless | 2.35 [1.90 to 2.90]

26. Secondary Outcome: Hill Coefficient (GAM) Derived From Statistical Analysis of the Relationship Between LAG3 Positive T Cell Levels in Blood and GSK2831781 Concentrations in Plasma (Part A and B)
Description: Blood samples were collected to measure LAG3 positive T cell levels. Plasma samples were collected to measure concentrations of GSK2831781 in plasma. The relationship between the pharmacodynamic measure (LAG3 positive T cell levels in blood) and plasma concentrations of GSK2831781 was described by an indirect response (Emax type) PK/PD model. The Hill coefficient GAM, a unitless parameter defining the steepness of the concentration-effect curve, was calculated by fitting the PK/PD model to all available data (Part A and Part B) of GSK2831781 concentrations in plasma and LAG3 positive T cells in blood. The model parameter; GAM is presented.
Time Frame: Up to Day 112
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Part A and Part B: All Participants
Number analyzed (Participants) | 28
Unitless | 0.0942 [0.0453 to 0.196]

27. Secondary Outcome: Part A: Number of Participants With Confirmed Positive Post-Baseline Anti-drug Antibody Result
Description: Serum samples were analyzed for the presence of anti-GSK2831781 antibodies using a validated immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'confirmed positive'. Number of participants with confirmed positive post-Baseline ADA result are presented.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants
Number analyzed (Participants) | 2 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0

28. Secondary Outcome: Part B: Number of Participants With Confirmed Positive Post-Baseline Anti-drug Antibody Result
Description: as for outcome 27
Time Frame: Up to Day 112
Population: Safety Population. Placebo arms across similar dosing strategies were combined in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
Number analyzed (Participants) | 4 | 8 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment (Day 1) up to Day 112 in Part A and in Part B
Description: SAEs and non-serious AEs were reported for the Safety Population which comprised of all randomized participants who received study intervention. Placebo arms across similar dosing strategies were combined in Part B.
Arm/Group | Part A: Placebo IV- Caucasian Participants | Part A: GSK2831781 450 mg IV- Caucasian Participants | Part A: Placebo IV- Japanese Participants | Part A: GSK2831781 450 mg IV- Japanese Participants | Part B: Placebo SC | Part B: GSK2831781 150 mg SC | Part B: GSK2831781 450 mg SC
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/2 | 0/6 | 0/4 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/2 | 0/6 | 0/4 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/2 | 5/6 | 0/2 | 4/6 | 4/4 | 6/8 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo IV- Caucasian Participants (N=2) | Part A: GSK2831781 450 mg IV- Caucasian Participants (N=6) | Part A: Placebo IV- Japanese Participants (N=2) | Part A: GSK2831781 450 mg IV- Japanese Participants (N=6) | Part B: Placebo SC (N=4) | Part B: GSK2831781 150 mg SC (N=8) | Part B: GSK2831781 450 mg SC (N=8)
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo IV- Caucasian Participants (N=2) | Part A: GSK2831781 450 mg IV- Caucasian Participants (N=6) | Part A: Placebo IV- Japanese Participants (N=2) | Part A: GSK2831781 450 mg IV- Japanese Participants (N=6) | Part B: Placebo SC (N=4) | Part B: GSK2831781 150 mg SC (N=8) | Part B: GSK2831781 450 mg SC (N=8)
Injection site bruising (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03965533/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03965533/SAP_001.pdf